CLINICAL TRIAL: NCT00235963
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Simvastatin on Subarachnoid Hemorrhage-Induced Vasospasm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Cenk Ayata, MD, Massachusetts General Hopital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2002-P-000215
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Subarachnoid Hemorrhage; Delayed Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
To determine whether HMG-CoA reductase inhibitor simvastatin prevents or ameliorates subarachnoid hemorrhage-induced delayed vasospasm and its ischemic consequences.

DETAILED DESCRIPTION:
The mortality rate of aneurysmal subarachnoid hemorrhage (SAH) approaches 50% within the 1st 24 hours of ictus. Patients who survive can subsequently develop a progressive vasospasm of large cerebral arteries, which is a major cause of morbidity and mortality. Vasospasm can be of varying severity, and only a small portion of patients with vasospasm develop clinical signs or symptoms. Patients with severe vasospasm are prone to develop ischemic deficits, which, if untreated, will progress into ischemic infarcts.

The mechanisms of vasospasm have been subject to intense investigation. Nitric oxide (NO)-cGMP system has attracted particular attention. Under normal physiological conditions, NO synthesized by endothelia NO synthase (eNOS) stimulates vascular smooth muscle cGMP production, which in turn causes smooth muscle relaxation. Vasospasm impairs endothelium-dependent dilations, suggesting that SAH induces a state of NO deficiency within cerebral arteries.

There are several potential mechanisms of such an NO deficiency. Hemoglobin is a potent scavenger of NO, and when applied extraluminal it binds NO and inhibits its action. Presence of perivascular hemoglobin may contribute to development of vasospasm by reducing the availability of NO. It has been shown that adventitial applied hemoglobin can inhibit basal NO activity and that in vivo adventitial exposure to whole blood leads to a reduction in basal cGMP levels in association with vasospasm of cerebral arteries. Similarly, superoxide also reacts with NO and acts as an NO scavenger. Superoxide production is increased after SAH, which may in part be responsible for inhibition of NO-dependent vasodilation. Free radical scavengers and manipulations to reduce free radical formation reduce vasospasm after SAH.

NOS is constitutively expressed in endothelium and adventitial perivascular nerve fibers. SAH-induced vasospasm in monkeys has been associated with diminished constitutive NOS immunoreactivity in the perivascular nerves around the spastic arteries. Endothelial NOS mRNA has also been decreased in monkey cerebral arteries 7d after SAH. Therefore, data suggest that there is a relative reduction in NO synthesis after SAH, in addition to increased breakdown.

In summary, the reduction in NO tonus around the cerebral arteries induced by decreased expression of endothelial NOS as well as increased NO scavenger substances in the subarachnoid space, and a relative resistance to NO-induced vasodilation in SAH appears to be one of the key events in the development of vasospasm. Therefore, therapeutic interventions that enhance endothelial NO production may compensate for these changes and reverse or reduce vasospasm.

Statins are FDA approved mainly as antihyperlipidemics, and they effectively reduce the risk of stroke and myocardial infarction. Simvastatin is also FDA-approved for stroke prevention. The risk reduction, however, is not correlated with the degree of lipid reduction, and is seen even in individuals with normal lipid levels. Statins are also cerebroprotective in stroke. They enhance endothelium-dependent relaxations, augment cerebral blood flow, reduce cerebral infarct size, and improve neurological outcome of stroke in normocholesterolemic animals. Their protective effects are independent of lipid reduction. Most importantly, statins upregulate endothelial NOS expression. This in turn improves cerebral blood flow and reduces infarct size in experimental models. In addition, statin treatment enhances endothelial fibrinolytic action, and inhibits platelet aggregation. Therefore, statins are excellent candidates to test on SAH-induced vasospasm.

This study has a randomized, double blind, placebo-controlled design. The anticipated enrollment is 104 patients, 52 in simvastatin, and 52 in placebo group, all recruited and studied at MGH. Assuming a difference of 27% or more, the power of this study is 88%, and alpha=0.05.

Inclusion and exclusion criteria are summarized below. Once enrolled, patients are randomized by Research Pharmacy staff to receive either placebo, or simvastatin 80 mg once every day, the highest clinically used dose of simvastatin. We chose this dose to maximize the effect on endothelium, which has been dose dependent in experimental studies. The study investigators are blinded to the treatment group. Patients are followed prospectively and receive standard aneurysmal subarachnoid hemorrhage care. The data collected pertains to development of vasospasm, and hence involves daily vital signs, neurologic examination, and routine neuroimaging. The development of vasospasm is determined based on daily transcranial Doppler studies, conventional angiography (routinely done within 7 days after subarachnoid hemorrhage as standard of care), and neurologic examination. Liver function tests along with total CPK are checked on admission and once a week for as long as the drug is continued, to screen for potential toxicity from the medication. Medication is discontinued if CPK or liver enzymes are elevated by more than 3 times the upper limit of normal range. CPK elevations due to surgical or percutaneous/endovascular interventions, or from cardiac sources (i.e. accompanied by troponin elevation with or without ECG changes), are not considered as indications for drug discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Aneurysmal subarachnoid hemorrhage, Fisher Grade III.
2. Patient or spouse or first degree relative able to give informed consent
3. Age greater then 18
4. Aneurysm secured surgically, or via endovascular technique
5. Subject seen within 96 hours of bleeding

Exclusion Criteria:

1. Contraindication for the use of simvastatin
2. Hunt-Hess Grade V
3. Initial intracranial pressure over 30 cm H2O and sustained for more then 30 minutes
4. Patient already on an HMG CoA-reductase inhibitor.
5. Patients with severe chronic renal failure (creatinine >3 and/or BUN >40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104
Dates: Start 2002-12; Primary Completion 2006-01 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Ayata, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chou SH, Smith EE, Badjatia N, Nogueira RG, Sims JR 2nd, Ogilvy CS, Rordorf GA, Ayata C. A randomized, double-blind, placebo-controlled pilot study of simvastatin in aneurysmal subarachnoid hemorrhage. Stroke. 2008 Oct;39(10):2891-3. doi: 10.1161/STROKEAHA.107.505875. Epub 2008 Jul 24. PMID 18658043